CLINICAL TRIAL: NCT02921724
Title: Participatory Research for Fine-tuning of a 2.0 System to Optimise Home Management of Oral Cancer Therapies.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRST100.18
Record Dates: First submitted 2016-09-26; First posted 2016-10-03 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Cancer; Oral Drug Administration
Keywords: cancer; oral drug; sunitinib; capecitabine; mobile app
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cancer patients undergoing oral therapy (Experimental): At the time of therapy prescription, patients candidate for oral therapy with capecitabine or sunitinib will be provided with informations on the side-effects of therapy and on the use and functions of the mobile diary app TreC-Onco. Patients are required to manually insert data into the mobile diary app at least once a day. Patients will be visited every 6 weeks. During the visit, the clinician will compare adherence and toxicity data entered into the mobile diary app with those directly reported by the patient and by drug accountability.
  Interventions: Device: TreC-Onco

INTERVENTIONS:
Device: TreC-Onco — TreC-Onco is composed of two tools aimed at supporting patient self-care and health professional monitoring and intervention:
  1. Mobile diary app. This is an Android app (for Android version 2.2 and higher) that allows patients to record parameters related to their health state (e.g. medications; blood pressure, weight, fever; side-effects or other symptoms) through a mobile device. Data are stored in a central database and are made available in real time to health professionals through a web dashboard on the TreC server or through a tablet app.
  2. Web dashboard. Through this, oncologists can check patient data, monitoring their side-effects and adherence to prescriptions. The Dashboard is optimized for the Firefox browser in version 7 or higher.

SUMMARY:
This is a prospective testing-validation, interventional, non-pharmacological study on a new app for oral anticancer therapy management.

A total of 80 patients will be considered: 20 evaluable patients in the training step; 60 patients in the validation step. In the training step will be considered evaluable the patients with: at least 6 weeks of treatment; visit at 6 weeks after the start of treatment performed and questionnaires self-administered.

Patients will be visited every 6 weeks. In the training step, patients will remain under observation for a minimum of 6 weeks, until change of therapy (due to progression of disease, unacceptable toxicity, death, discontinuation) or for a maximum of 12 weeks. Patients enrolled in the validation step will remain under observation until change of therapy (due to progression of disease, unacceptable toxicity, death, discontinuation) or for a maximum of 24 weeks.

The objective of this study is to assess the capability of a newly developed interactive health care application to support patients and health professionals in the shared management of oral anticancer therapies, improving adherence, preventing complications at home, toxicities, improper treatment reductions or interruptions, emergency accesses and to assess the system usability and acceptability by patients and health professionals, integration in the hospital workflow, monitoring over time patient perceived levels of quality of care, quality of life, social support, anxiety, and self-care capability.

DETAILED DESCRIPTION:
This is a prospective, interventional, non pharmacological study for testing-validation of a new app for optimising home management of oral therapies for cancer treatment.

All patients will be treated according to the local clinical practice. Enrolment period: 8 (training step) + 12 (validation step) months. Total duration of the study: 36 months. This is a multicenter study. Objective of the study is to assess the capability of a newly developed interactive health care application to support patients and health professionals in the shared management of oral anticancer therapies, and to assess the system usability and acceptability by patients and health professionals.

Eligible patients must meet the following criteria:

* adult 18-75 years old;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
* candidate for treatment with capecitabine or sunitinib as monotherapy (adjuvant and advanced settings allowed);
* sufficient ability to manage mobile devices after basic training course held at baseline;
* clear understanding of the Italian language;
* written informed consent.

Health professionals and patients define the items of the system through participatory design techniques (e.g. focus group sessions, joint review).

To define whether the system is capable of monitoring patient adherence, the number of pills counted by the system (self-reported by the patient at home) will be compared with that counted by the physician as residual pills returned by the patient at the hospital visit. A difference in the number of pills within +/- 10% will be considered acceptable. A comparison of type and grade of toxicity will be made between the adverse events indicated by the system and those reported by the patient at the clinical visit. The quality of the system will be considered adequate if all the grade 3 and at least 80% of the grade 2 or more toxicity data reported by the patient at the time of the visit is recorded in the app.

To investigate system usability and acceptability, Functional Assessment of Cancer Therapy-General (FACT-G) and Hospital Anxiety and Depression Scale (HADS) questionnaires will be used. Scores will be subdivided into different subscales and analyzed using the Wilcoxon rank-sum test. Two new questionnaires have been developed and will be used to evaluate patient expectations of the system, and system acceptability + patient-doctor communication. An internationally validated questionnaire translated into Italian on system usability (SUS) will be also administered at the end of observation. Conversational interviews will be audio-recorded, transcribed and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* ECOG-Performance Status (PS) less or equal to 1;
* life expectancy > 12 weeks;
* candidate for treatment with capecitabine or sunitinib as monotherapy (adjuvant and advanced settings allowed);
* clear understanding of the Italian language;
* subjects who are, in the opinion of the Investigator, able to understand this study, to cooperate with the study procedures and able to manage mobile devices after basic training course held at baseline;
* written informed consent

Exclusion Criteria:

* Patients receiving also intravenous anticancer treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Drug accountability comparison | 3 years
  the number of pills counted by the system (self-reported by the patient at home) will be compared with that counted by the physician as residual pills returned by the patient at the hospital visit. A difference in the number of pills within +/- 10% will be considered acceptable.
Toxicity reporting comparison | 3 years
  A comparison of type and grade of toxicity will be made between the adverse events indicated by the system and those reported by the patient/detected by the doctor at the clinical visit. The quality of the system will be considered adequate if all the grade 3 and at least 80% of the grade 2 toxicity data reported by the patient at the time of the visit is recorded in the app. A comparison will be made between the adverse event start time reported by the system and the time of data-entry by the patient into the system.

SECONDARY OUTCOMES:
System acceptability: HADS questionaire | 3 years
  HADS questionaire will be analyzed using the Wilcoxon rank-sum test
System acceptability: FACT-B questionaire | 3 years
  FACT-B questionaire will be analyzed using the Wilcoxon rank-sum test
System usability: system usability scale (SUS) questionaire | 3 years
  system usability scale (SUS) will be analyzed using the Wilcoxon rank-sum test
System acceptability by the Q-pre questionaire | 3 years
  System acceptability by the Q-pre questionaire using content and template qualitative sociological analysis
System acceptability by the Q-post questionaire | 3 years
  System acceptability by the Q-post questionaire using content and template qualitative sociological analysis
System acceptability by semi-structured interviews | 3 years
  System acceptability by semi-structured interviews using content and template qualitative sociological analysis

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Passardi, MD, Study Chair — IRST IRCCS, Meldola (FC)
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Bergamo
  - Irst-Irccs, Meldola (FC)
  - Azienda Provinciale per i Servizi Sanitari della Provincia Autonoma di Trento, Trento

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Passardi A, Foca F, Caffo O, Tondini CA, Zambelli A, Vespignani R, Bartolini G, Sullo FG, Andreis D, Dianti M, Eccher C, Piras EM, Forti S. A Remote Monitoring System to Optimize the Home Management of Oral Anticancer Therapies (ONCO-TreC): Prospective Training-Validation Trial. J Med Internet Res. 2022 Jan 26;24(1):e27349. doi: 10.2196/27349. PMID 35080505
- [Derived] Passardi A, Rizzo M, Maines F, Tondini C, Zambelli A, Vespignani R, Andreis D, Massa I, Dianti M, Forti S, Piras EM, Eccher C. Optimisation and validation of a remote monitoring system (Onco-TreC) for home-based management of oral anticancer therapies: an Italian multicentre feasibility study. BMJ Open. 2017 May 29;7(5):e014617. doi: 10.1136/bmjopen-2016-014617. PMID 28554917